CLINICAL TRIAL: NCT01202045
Title: Stress Echocardiography in the Detection of Pulmonary Arterial Hypertension in Systemic Sclerosis Patients With Indirect Signs of Pulmonary Arterial Hypertension
Brief Title: Stress Echocardiography in the Detection of Pulmonary Arterial Hypertension in Systemic Sclerosis Patients
Status: Withdrawn | Type: Observational
Sponsor: Paul Farand (Other)
Responsible Party: Sponsor-Investigator, Paul Farand, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Other Study IDs: Projet # 10-111
Record Dates: First submitted 2010-09-10; First posted 2010-09-15 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Scleroderma, Systemic; Hypertension, Pulmonary
Keywords: Echocardiography, Stress; right heart catheterization
MeSH Terms: conditions — Scleroderma, Systemic; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- systemic sclerosis patients: Every patient will have a rest echocardiography, a stress echocardiography, a right heart catheterization, a blood specimen, and a pulmonary function test.

SUMMARY:
The purpose of this study is to assess the value in terms of sensitivity, specificity and likelihood ratio of the stress echocardiography in the screening of pulmonary arterial hypertension in patients with systemic sclerosis and indirect signs of pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Pulmonary artery catheterization (rest and exertion) and treadmill stress echocardiography will be done to all patients of the study.

ELIGIBILITY:
Inclusion Criteria:

* At least one of the prespecified indirect sign of pulmonary arterial hypertension
* Able to exercise on treadmill

Exclusion Criteria:

* left ventricular dysfunction at rest
* Absence of pulmonary regurgitant flow
* Pregnancy or breastfeeding
* Smoking with > 60 pack-year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systemic slerosis patients with indirect signs of arterial pulmonary hypertension:
  * Effort dyspnea (NYHA >= 2/4)
  * DLCO < 60%
  * FVC% / DLCO% > 1.6
  * SPAP > 40 mmhg and < 55 mmhg
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Correlation of a 20 mmhg increase in the pulmonary artery pressures (PAP) during stress echocardiography and PAP using right heart catheterization. | 5 years
  Every patient will have both procedures; stress echocardiography and right heart catheterization. A positive stress echocardiography is defined as >= 20 mmhg increase in the systolic pulmonary artery pressure (SPAP) (between rest and stress) or an absolute value >= 55 mmhg. A positive right heart catheterization at rest is defined as a PAPm >25mmhg, wedge < 18 and pulmonary vascular resistances >3 wood units. Stress catheterization will also be perform and is defined as a PAPm > 30mmhg and wedge <18 mm hg.

SECONDARY OUTCOMES:
Correlation of a 20 mmhg increase in the PAP during stress echocardiography and elevated NT-proBNP. | 5 years
Function of the left ventricle (left ventricular ejection fraction) at rest and at stress. | Follow up every year X 5
  We hypothesize that patients who do not increase their left ventricular ejection fraction at stress have a worst clinical outcome in the follow up.
Diastolic function at rest and at stress | follow up every year X 5
  We hypothesize that patients with diastolic dysfunction manifesting at stress have a worst clinical outcome in the follow up.
Function of the right ventricle | Follow up every year X 5
  We hypothesise that in patients with or without pulmonary hypertension, right ventricular dysfunction is associated with a worse clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Paul Farand, md, msc, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada